CLINICAL TRIAL: NCT01751529
Title: LCCC 1219: A Prospective Pilot Study Evaluating Renal Lesions Through Contrast-enhanced US in Patients With Renal Cancer and in Those With a Risk Factor for Renal Malignancy
Brief Title: Open-label Pilot Evaluating Renal Lesions w/ Contrast-enhaced US in Patients w/ Renal Cancer
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC 1219
Record Dates: First submitted 2012-12-13; First posted 2012-12-18 (Estimated); Last update posted 2017-03-17 (Actual); Status verified 2017-03

CONDITIONS: Kidney Cancer
Keywords: renal malignancy; Pilot Study; LCCC 1219; UNC Lineberger; kidney cancer; contrast-enhanced ultrasound; ultrasound
MeSH Terms: conditions — Kidney Neoplasms | interventions — perflutren

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Contrast-enhanced Ultrasound (Experimental)
  Interventions: Procedure: Contrast-enhanced Ultrasound; Drug: Perflutren lipid

INTERVENTIONS:
Procedure: Contrast-enhanced Ultrasound — All patients will undergo a contrast-enhanced ultrasound prior to planned resection or ablative therapy or as part of routine screening for kidney cancer.
  Other Names: Contrast-enhanced US
Drug: Perflutren lipid — All patients will receive a contrast-enhanced ultrasound using microbubble contrast agent (perflutren lipid; Definity®) prior to planned resection or ablative therapy or as part of routine screening for kidney cancer.
  Other Names: Definity®

SUMMARY:
This prospective pilot study is designed to evaluate the accuracy of contrast-enhanced ultrasound when used to evaluate renal lesions in two different populations; patients with known renal tumors (Cohort 1) and patients with a risk factor for renal malignancy in whom their screening ultrasound shows an indeterminate or possibly malignant renal mass (Cohort 2).

DETAILED DESCRIPTION:
This prospective pilot study is designed to evaluate the accuracy of contrast-enhanced ultrasound using microbubble contrast agent (perflutren lipid; Definity®) when used to evaluate renal lesions in two different populations; patients with known renal tumors (Cohort 1) and patients with a risk factor for renal malignancy in whom their screening ultrasound shows an indeterminate or possibly malignant renal mass (Cohort 2).

ELIGIBILITY:
Inclusion Criteria:

1. Able to provide written informed consent
2. Willing to comply with protocol requirements
3. At least 18 years of age
4. Cohort 1:

   * Be eligible for radical or partial nephrectomy or ablative therapy based upon at least one renal lesion identified during previous contrast enhanced CT or MR.

   OR
5. Cohort 2:

   * High risk group (patient recommended for routine surveillance screening for renal malignancy)
   * Have at least one kidney lesion identified but incompletely characterized on a screening US, CT, or MR exam

Exclusion Criteria:

1. Critically ill or medically unstable and whose critical course during the observation period would be unpredictable (e.g., chronic obstructive pulmonary disease (COPD) requiring oxygen)
2. Known hypersensitivity to sulfur hexafluoride or to any component of perflutren lipid (Definity®)
3. Right to left shunt, severe pulmonary hypertension (Pulmonary artery pressure >90mmHg), or adult respiratory distress syndrome
4. Active cardiac disease including any of the following:

   * Severe congestive heart failure (class IV in accordance with the classification of the New York Heart Association)
   * Unstable angina.
   * Severe arrhythmia (i.e. ventricular tachycardia, flutter fibrillation; ventricular premature complexes occurring close to the preceding T-wave, multifocal complexes).
   * Myocardial infarction within 14 days prior to the date of proposed Definity® administration.
   * Uncontrolled systemic hypertension (Blood pressure: systolic blood pressure (BP) >150 mm Hg and/or diastolic BP >90 mm Hg despite optimal medical management not controllable by medication to achieve BP <15/90)
5. Is in an intensive care setting
6. Has an unstable neurological disease (e.g recent stroke or TIA symptoms (<3 months)) cerebrovascular accident (including transient ischemic attacks (TIAs) within the 3 months before signing of informed consent
7. Undergone an invasive procedure on kidney lesion (e.g. tissue biopsy, surgery, nonsurgical cytoreductive procedure) in-between identification of lesion via US without contrast and perflutren lipid administration
8. Has previously been entered into this study or has received an investigational drug within the 30 days prior to admission into this study
9. Has any other medical condition or other circumstances that would significantly decrease the chances of obtaining reliable data or of achieving the study objectives such as:

   * Mental illness
   * Drug abuse
10. Female patient who is pregnant or lactating (the possibility of pregnancy has to be excluded by negative serum or urine B-HCG results, obtained within 24 hours before the perflutren lipid administration, or on the basis of patient history, e.g.: tubal ligation, hysterectomy or a minimum of 1 year without menses).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2013-05; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of using contrast-enhanced ultrasound in diagnosing renal malignancy in patients with known renal disease (Cohort 1) and in patients with a risk factor for renal malignancy diagnosed with suspicious or indeterminate lesions (Cohort 2) | 12 months
  Primary analyses will include 1) estimating the sensitivity of contrast enhanced ultrasound in Cohort 1 using the pathological outcome or biopsy result from ablative therapy as gold standard and 2) estimating sensitivity in Cohort 2 using pathology and follow-up results as gold standard (when tissue biopsy is not indicated nor surgery planned the truth standard diagnosis will be based on 12 month follow-up data of disease status). Exact 95% confidence intervals for sensitivity estimate will be reported.

SECONDARY OUTCOMES:
Feasibility of comparing the sensitivity and specificity of contrast enhanced ultrasound to traditional imaging techniques (CT and MRI) in detecting renal lesions in patients already diagnosed with a renal malignancy | 12 months
  The estimates obtained in Cohort 1 will be compared to the published figures of the conventional CT and MRI method. For Cohort 2 patients who undergo surgery, the percentage of subjects who are correctly diagnosed (benign and malignancy) will be reported along with exact 95% CI. Frequency tables will be used to describe associations. Appropriate descriptive summary statistics such as mean, median and standard deviation of tumor measurement will be provided to quantify and characterize renal masses.

CONTACTS AND LOCATIONS:
Overall Officials: Kimryn Rathmell, MD, Principal Investigator — University of North Carolina; Wui Chong, MBBS, FRCR, Principal Investigator — University of North Carolina
Locations (1):
- Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Chang EH, Chong WK, Kasoji SK, Fielding JR, Altun E, Mullin LB, Kim JI, Fine JP, Dayton PA, Rathmell WK. Diagnostic accuracy of contrast-enhanced ultrasound for characterization of kidney lesions in patients with and without chronic kidney disease. BMC Nephrol. 2017 Aug 9;18(1):266. doi: 10.1186/s12882-017-0681-8. PMID 28793871
- See also: Lineberger Comprehensive Cancer Center website — http://unclineberger.org/
- See also: National Cancer Institute (NCI) website — http://www.cancer.gov/